CLINICAL TRIAL: NCT06006221
Title: The Effect of Qigong Intervention on State Anxiety Levels of Inpatiens in Psychiatric Wards: A Randomized Controlled Study
Brief Title: Qigong Intervention and State Anxiety Levels of Inpatiens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emel Erdeniz Güreş (Other)
Responsible Party: Sponsor-Investigator, Emel Erdeniz Güreş, Research Assistant, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0000000339492770
Record Dates: First submitted 2023-08-14; First posted 2023-08-23 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Psychiatric Disorder
Keywords: psychiatric service,Qi Gong, nursing
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After the morning meeting, the initiative group will be given 40 minutes of Qigong relaxation exercise.
  Interventions: Behavioral: Qi-gong relaxation exercise
- control group (No Intervention): No application will be made to the control group. The control group will continue their routine treatment in the clinic.

INTERVENTIONS:
Behavioral: Qi-gong relaxation exercise — Qi-gong relaxation exercise is a mindfulness-based exercise and is a type of exercise that consists of breathing-compatible body movements and relaxation used to relax the body and mind, reduce stress, distract attention from negative thoughts, accelerate blood flow, and improve emotions.
  Arms: experimental group

SUMMARY:
The aim of the study, which aimed to examine the effect of the Qigong relaxation exercise applied in psychiatry clinics on the level of anxiety, was planned as randomized controlled. Individuals will be divided into intervention and control groups. Before the application, the Personal Information Form and STAI Form I scale will be applied to the patients in the Intervention and Control group. Patients in the intervention group are expected to answer the STAI Form I scale after qigong relaxation exercises. It planned to apply the same forms as planned in the intervention group without any application in the control group. Personal Information Form and STAI Form I Scale will be filled by the patients in the form of self-report.

DETAILED DESCRIPTION:
Anxiety is one of the most common and compelling symptoms in individuals receiving treatment in psychiatry clinics. The issue of managing anxiety is very important in psychiatry clinics. Various pharmacological, physical, and therapeutic methods are applied to reduce and manage these symptoms. In addition to pharmacologically applied medical treatment, non-drug applications used as supportive are recommended in terms of reducing the symptoms of the disease and increasing the quality of life of the individual. These non-drug methods are; aromatherapy, physical exercise, light therapy, and music therapy. physical exercise; It is defined as planned, structured, repetitive movements to promote or maintain physical and mental health. Aerobics (brisk walking, dancing, cycling), endurance and resistance (squeezing rubber balls using elastic resistance bands and lifting weights), and flexibility and balance exercises (qigong, yoga, and pilates) are examples of physical exercises. In the literature, the effect of Qigong practices on anxiety in many patient groups has been examined, but no study has been found on the effect of Qigong relaxation exercises on the level of anxiety in inpatient psychiatric patients. Therefore, this study aims to examine the effect of Qigong relaxation exercises applied in the psychiatry clinic on the anxiety level of patients. Patients will be divided into intervention and control groups in a randomized controlled manner. After obtaining ethics committee approvals for the intervention group, clinics will be informed about the Qigong relaxation exercises study and it will be planned to place this study in the daytime program with the clinicians. The most appropriate time for patients to practice qigong relaxation exercises was determined after the morning meeting. No qigong exercise will be performed for the control group. Before the application, the Personal Information Form, STAI Form I, will be applied to the patients in the Intervention and Control group. Patients in the intervention group are expected to answer the STAI Form I scale after qigong relaxation exercises. It planned to apply the same forms as planned in the intervention group without any application in the control group. Personal Information Form and STAI Form I Scale will be filled by the patients in the form of self-report. The practice of the qigong relaxation exercise will take place after the good morning meetings. Qigong relaxation exercise is a mindfulness-based exercise and is a type of exercise consisting of body movements and relaxation in harmony with breathing used to relax the body and mind, reduce stress, distract attention from negative thoughts, accelerate blood flow, and improve emotions. It is planned to apply this exercise once for 40 minutes to the patients included in the intervention group as a group activity by researchers trained on this subject.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is literate and has no communication barriers
2. Being an inpatient in the psychiatry clinic
3. Being over 18 years old
4. The patient has been oriented to the service (at least 24 hours have passed since his hospitalization)
5. Regular participation in qigong practice

Exclusion Criteria:

1. The patient has communication difficulties
2. Having acute psychotic symptoms
3. Patients receiving anxiolytic therapy

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | three month
  The personal information form was created by the researchers and includes demographic information and information about the disease. Demographic information consists of seven questions about age, gender, marital status, educational status, employment status, with whom she lives and whether she has a visitor in the clinic. Information about the disease; It consists of eight questions about psychiatric diagnosis, symptoms of hospitalization, duration of illness, number of hospitalizations, drugs used, whether ECT was applied, whether chemical and isolation practices were applied.
STAI Anxiety Scale I | three month
  Developed by Spielberger in 1970, its Turkish version was developed by Öner N et al. The validity and reliability study was carried out by adapting it. It is a likert type scale that measures state anxiety levels with 20 questions. Anxiety level is scored as "(1) not at all, (2) a little, (3) a lot, and (4) completely" in STAI-I. Direct statements on the scale, negative emotions; reversed expressions express positive emotions. Two separate total score weights are calculated for each of the direct and reversed statements. The total score for the reverse statements is subtracted from the total score for the direct statements. A predetermined and unchanging value is added to this number. A constant value of 50 was added to the number obtained for STAI-I. The most recent value indicates the individual's anxiety score. The scores obtained from the scale range from 20 to 80. A high score indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AS, Cheung MC, Sze SL, Leung WW, Shi D. Shaolin dan tian breathing fosters relaxed and attentive mind: a randomized controlled neuro-electrophysiological study. Evid Based Complement Alternat Med. 2011;2011:180704. doi: 10.1155/2011/180704. Epub 2010 Sep 22. PMID 20976126
- [Background] Abbott R, Lavretsky H. Tai Chi and Qigong for the treatment and prevention of mental disorders. Psychiatr Clin North Am. 2013 Mar;36(1):109-19. doi: 10.1016/j.psc.2013.01.011. PMID 23538081
- [Background] Wang CW, Chan CL, Ho RT, Tsang HW, Chan CH, Ng SM. The effect of qigong on depressive and anxiety symptoms: a systematic review and meta-analysis of randomized controlled trials. Evid Based Complement Alternat Med. 2013;2013:716094. doi: 10.1155/2013/716094. Epub 2013 May 20. PMID 23762156
- [Background] Wang CW, Chan CH, Ho RT, Chan JS, Ng SM, Chan CL. Managing stress and anxiety through qigong exercise in healthy adults: a systematic review and meta-analysis of randomized controlled trials. BMC Complement Altern Med. 2014 Jan 9;14:8. doi: 10.1186/1472-6882-14-8. PMID 24400778
- [Background] Chang PS, Knobf MT, Oh B, Funk M. Physical and psychological effects of Qigong exercise in community-dwelling older adults: An exploratory study. Geriatr Nurs. 2018 Jan-Feb;39(1):88-94. doi: 10.1016/j.gerinurse.2017.07.004. Epub 2017 Aug 17. PMID 28822591
- [Background] Guo Y, Xu M, Zhang J, Hu Q, Zhou Z, Wei Z, Yan J, Chen Y, Lyu J, Shao X, Wang Y, Guo J, Wei Y. The effect of Three-Circle Post Standing (Zhanzhuang) Qigong on the physical and psychological well-being of college students: Study protocol for a randomized controlled trial. Medicine (Baltimore). 2018 Sep;97(38):e12323. doi: 10.1097/MD.0000000000012323. PMID 30235685
- [Background] Oh B, Choi SM, Inamori A, Rosenthal D, Yeung A. Effects of qigong on depression: a systemic review. Evid Based Complement Alternat Med. 2013;2013:134737. doi: 10.1155/2013/134737. Epub 2013 Mar 4. PMID 23533461
- [Background] Chen CH, Hung KS, Chung YC, Yeh ML. Mind-body interactive qigong improves physical and mental aspects of quality of life in inpatients with stroke: A randomized control study. Eur J Cardiovasc Nurs. 2019 Dec;18(8):658-666. doi: 10.1177/1474515119860232. Epub 2019 Jun 23. PMID 31232097
- [Background] Xu S, Zhang D, He Q, Ma C, Ye S, Ge L, Zhang L, Liu W, Chen Z, Zhou L. Efficacy of Liuzijue Qigong in patients with chronic obstructive pulmonary disease: A systematic review and meta-analysis. Complement Ther Med. 2022 May;65:102809. doi: 10.1016/j.ctim.2022.102809. Epub 2022 Jan 29. PMID 35093513
- [Background] Molassiotis A, Vu DV, Ching SSY. The Effectiveness of Qigong in Managing a Cluster of Symptoms (Breathlessness-Fatigue-Anxiety) in Patients with Lung Cancer: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211008253. doi: 10.1177/15347354211008253. PMID 33847150
- [Background] Roswiyani R, Hiew CH, Witteman CLM, Satiadarma MP, Spijker J. Art activities and qigong exercise for the well-being of older adults in nursing homes in Indonesia: a randomized controlled trial. Aging Ment Health. 2020 Oct;24(10):1569-1578. doi: 10.1080/13607863.2019.1617239. Epub 2019 May 30. PMID 31146543
- [Background] Sultana M, Bryant D, Orange JB, Beedie T, Montero-Odasso M. Effect of Wii Fit(c) Exercise on Balance of Older Adults with Neurocognitive Disorders: A Meta-Analysis. J Alzheimers Dis. 2020;75(3):817-826. doi: 10.3233/JAD-191301. PMID 32310168
- [Background] Park J, Howard H, Tolea MI, Galvin JE. Perceived Benefits of Using Nonpharmacological Interventions in Older Adults With Alzheimer's Disease or Dementia With Lewy Bodies. J Gerontol Nurs. 2020 Jan 1;46(1):37-46. doi: 10.3928/00989134-20191217-01. PMID 31895960
- [Background] Özmen, E.ve Taşkın E.O., Ruhsal Hastalıklara Yönelik Tutumların Ruh Sağlığı Hizmetlerine Etkisi Stigma Ruhsal Hastalıklara Yönelik Tutumlar ve Damgalama, İzmir, 2007.
- [Background] Kelleci M., Aydın D., Sabancıoğulları S., Doğan S. Hastanede Yatan Hastaların Bazı Tanı Gruplarına Göre Anksiyete ve Depresyon Düzeyleri,2009.
- [Background] Kurt E. M., Kannabis kullanım bozukluğu hastalarında gastrointestinal sistem (GİS) hormonları ile agresyon ve aşerme arasındaki İlişkinin İncelenmesi, Uzmanlık Tezi Sakarya Üniversitesi, 2020.
- [Background] Savaşan, A., ve Mete, L. (2018). Bir eğitim ve araştırma hastanesi psikiyatri kliniklerinde agresyonun ve kısıtlama yöntemlerinin incelenmesi. Klinik Psikiyatri Dergisi, 21(2), 130-136.
- [Background] Şahin M., Korku, Kaygı ve Kaygı (Anksiyete) Bozuklukları, Avrasya Sosyal ve Ekonomi Araştırmaları Dergisi, Cilt 6. Sayı S 117-135,2019.